CLINICAL TRIAL: NCT07390786
Title: Integration of a Behavioral Health Collaborative Care Model Into an ICU Recovery Clinic-Pilot for Families
Brief Title: Behavioral Health Collaborative Care Model in Post-ICU Clinic Family Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rita Bakhru, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00145594
Record Dates: First submitted 2026-01-12; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness Recovery; Behavioral Health Concerns; Anxiety; Depression - Major Depressive Disorder; PTSD; Critical Care, Intensive Care; PICS-F
Keywords: Critical Ilness; critical care recovery; Post-Intensive Care Syndrome; Post-ICU care; behavioral health; mental health; anxiety; depression; PTSD; PICS-F
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; postintensive care syndrome; Psychological Well-Being; Depression | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Attention Control.
- Interventional (Experimental)
  Interventions: Behavioral: Behavioral Treatment

INTERVENTIONS:
Behavioral: Behavioral Treatment — behavioral health collaborative care model in ICU recovery patients and families
  Arms: Interventional

SUMMARY:
This pilot study evaluates the feasibility and acceptability of implementing a Behavioral Health Collaborative Care Model (BH CoCM) for family members of ICU survivors. The intervention includes telehealth-enabled behavioral health assessments and access to the NeuroFlow platform. A subset of participants will undergo qualitative interviews.

DETAILED DESCRIPTION:
Patients seen in the MUSC ICU Recovery Clinic will be approached for consent for care through our Behavioral Health Collaborative Care Model. Patients and their families that consent will be randomized to an attention control group or an intervention group.

The intervention group will have access to NeuroFlow platform, which has been specifically designed to support delivery of a BH CoCM. They will utilize Neuroflow for 6 months. They will undergo assessments for anxiety, depression, post-traumatic stress The attention control group will undergo assessments for anxiety, depression, post-traumatic stress.

Investigators will look at changes over six months in intervention group compared to attention control group for patients in terms of symptoms of depression, anxiety, post-traumatic stress. Investigators will also look at adherence, BH CoCM implementation metrics, type and amount of guided content accessed in NeuroFlow. Investigators will perform qualitative surveys to understand better what patients thought about the intervention and ways in which it could be improved.

ELIGIBILITY:
Inclusion Criteria:

- Family member of ICU Recovery Clinic patient enrolled in parent BH CoCM study

Exclusion Criteria:

* Serious mental illness (e.g., schizophrenia, mania)
* Late-stage dementia or cognitive impairment
* Limited English proficiency
* No internet-enabled device
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Consent Rate | Baseline
  Investigators will assess the consent rate
Study Completion Rate | enrollment to 6 months
  We will assess the completion rate of all enrolled family members

SECONDARY OUTCOMES:
Monthly Completion Rate of PHQ9 (Patient Health Questionnaire 9) | Enrollment to 6 months
  Rate of completion of scheduled monthly assessment: PHQ9
Monthly Completion Rate of GAD 7 (General Anxiety Disorder 7) | baseline to 6 months
  Rate of completion of scheduled monthly assessment: GAD7
Monthly Completion Rate of PCL 5 (PTSD Checklist for DSM-5) | baseline to 6 months
  Rate of Completion of scheduled monthly assessment: PCL5

CONTACTS AND LOCATIONS:
Overall Officials: Rita Bakhru, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be used for future research without additional consent.